CLINICAL TRIAL: NCT04367064
Title: To Study the Clinical Characteristics and Treatment Outcome of COVID-19 Patients Admitted in Hospitals of Max Healthcare (SCOPe Study)
Acronym: SCOPe
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Max Healthcare Insititute Limited (Other)
Responsible Party: Sponsor
Other Study IDs: SCOPe/MHC/Covid-19/2020
Record Dates: First submitted 2020-04-26; First posted 2020-04-29 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: COVID

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study for Corona virus disease by the Max Healthcare.Corona virus 2019 disease (COVID-19) is a respiratory tract infectious disease caused by a newly emergent corona virus. This virus is linked to the same family of viruses as Severe Acute Respiratory Syndrome (SARS) and some types of common cold.

DETAILED DESCRIPTION:
In view of increasing cases in India and the possibility of the exponential rise of cases, study has been designed to observe the patient profile and outcomes for hospitalized positive Covid-19 patients that may help to understand the effectiveness of different treatment strategies. This is a retrospective and prospective, observational study based on collection of data related to COVID-19 admitted patients treated in the hospitals of Max Healthcare as per the standard treatment protocol and policy for COVID 19 at Max Healthcare.

Covid19 patients shall be approached at the time of admission for participation in this study. If the patient consents, the participating investigator or designated study personnel will collect the baseline demographic details of the patient, along with medical history; current disease status; current and previous treatment details; and the results of all the laboratory tests performed, as per the standard clinical practices. Daily follow up will be done on a structured case record form (CRF) till the discharge or death.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either sex aged ≥18 years
2. Patients who are Covid-19 positive
3. All patients with positive Corona virus infection admitted in the hospitals of Max Healthcare will be included in the study.

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the confirmed cases of COVID 19 getting treated at Max Super Speciality Hospital (DDF) as per the standard treatment protocol and policy for COVID 19.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-04-25 (Actual); Primary Completion 2020-11-25 (Estimated); Study Completion 2020-12-25 (Estimated)

PRIMARY OUTCOMES:
we will compare the clinical outcome of the COVID 19 patients with their age and gender | 3-4 months
  Collection of the baseline demographic details of the patient, along with medical history; current disease status; current and previous treatment details; and the results of all the laboratory tests performed, as per the standard clinical practices. All the data will be entered into Excel sheet, row wise for each patient. For studying the demographic profile, the age will be divided into standard 10-year intervals and percentages will be obtained for each sex and combined for males and females. This will be in addition to the mean and SD of age.

SECONDARY OUTCOMES:
we will compare the effect of different treatments given to the COVID 19 patients at Max Hospital | 3-4 months
  Daily follow up will be done on a structured case record form (CRF) till the discharge or death of the subject. Treatment-Related Adverse Events as Assessed by CTCAE v4.0 will be captured in CRF. Clinical profile and outcome will be analyzed separately for each treatment regimen after suitable grouping of the regimens. Statistical significance of the association of outcomes with the clinical profile and treatment regimens will be checked with chi-square test or Fisher exact test in case the numbers are small. Effectiveness of each regimen will also be checked for significance of difference with chi-square test. A P-value <0.05 will be considered statistically significant but the final conclusion will be based on corroborative evidence and factors such as clinical profile. SPSS 20 will be used for all the calculations.

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Budhiraja, MRCP, FACP, Principal Investigator — Max Healthcare
Locations (1):
- Max Super Speciality hospital, Saket (A unit of Devki Devi Foundation), New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing is undecided at this stage. We may, however, provide the data if requested.